CLINICAL TRIAL: NCT01490671
Title: Phase 2 Expanded Safety Study of Tenofovir Gel in Pregnancy
Brief Title: Evaluating the Safety of Tenofovir Vaginal Gel in HIV-Uninfected Pregnant Women
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MTN-019; 11839 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group 1a (tenofovir gel) (Experimental): Group 1a will include women with a gestational age range of 36 0/7 to 37 6/7 weeks; they will receive 1% tenofovir gel
  Interventions: Drug: 1% tenofovir gel
- Group 1b (placebo gel) (Placebo Comparator): Group 1b will include women with a gestational age range of 36 0/7 to 37 6/7 weeks; they will receive placebo gel.
  Interventions: Drug: Placebo gel
- Group 2a (tenofovir gel) (Experimental): Group 2a will include women with a gestational age range of 28 0/7 to 32 6/7 weeks; they will receive 1% tenofovir gel.
  Interventions: Drug: 1% tenofovir gel
- Group 2b (placebo gel) (Placebo Comparator): Group 2b will include women with a gestational age range of 28 0/7 to 32 6/7 weeks; they will receive placebo gel.
  Interventions: Drug: Placebo gel
- Group 3a (tenofovir gel) (Experimental): Group 3a will include women with a gestational age range of 20 0/7 to 24 6/7 weeks; they will receive 1% tenofovir gel.
  Interventions: Drug: 1% tenofovir gel
- Group 3b (placebo gel) (Placebo Comparator): Group 3b will include women with a gestational age range of 20 0/7 to 24 6/7 weeks; they will receive placebo gel.
  Interventions: Drug: Placebo gel
- Group 4a (tenofovir gel) (Experimental): Group 4a will include women with a gestational age range of 12 0/7 to 16 6/7 weeks; they will receive 1% tenofovir gel.
  Interventions: Drug: 1% tenofovir gel
- Group 4b (placebo gel) (Placebo Comparator): Group 4b will include women with a gestational age range of 12 0/7 to 16 6/7 weeks; they will receive placebo gel.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: 1% tenofovir gel — One applicator of 1% tenofovir gel will be inserted by the participant into the vagina once each day for 28 days or until delivery, whichever comes first
  Arms: Group 1a (tenofovir gel); Group 2a (tenofovir gel); Group 3a (tenofovir gel); Group 4a (tenofovir gel)
Drug: Placebo gel — One applicator of placebo gel will be inserted by the participant into the vagina once each day for 28 days or until delivery, whichever comes first
  Arms: Group 1b (placebo gel); Group 2b (placebo gel); Group 3b (placebo gel); Group 4b (placebo gel)

SUMMARY:
Preliminary research has shown that a vaginal gel containing the antiretroviral (ARV) drug tenofovir may reduce the risk of HIV infection in women when used near the time of sexual intercourse. This study will evaluate the safety of 1% tenofovir gel in HIV-uninfected pregnant women and their newborns when the gel is used once a day for a period of 28 days at a designated time during pregnancy.

DETAILED DESCRIPTION:
Pregnant women often maintain sexual activity, and research has shown that they may have a greater risk of acquiring HIV infection during pregnancy. Preliminary research has suggested that tenofovir 1% gel, a vaginal microbicide, may reduce the risk of HIV infection for women when it is applied at the time of sexual intercourse. However, safety data on the use of tenofovir 1% gel during pregnancy are limited. This study will enroll pregnant women who will use tenofovir 1% gel on a daily basis for 28 consecutive days during their pregnancy, which is a longer period of use than has been studied previously. The purpose of this study is to evaluate the safety of 1% tenofovir gel in HIV-uninfected pregnant women when used during the late first trimester and second trimester of pregnancy.

Participants will be healthy, HIV-uninfected pregnant women and will be randomly assigned to use either 1% tenofovir gel or placebo gel once a day for 28 days or until delivery, whichever comes first. Participants will be further divided into four groups of varying gestational age ranges. These groups will be filled sequentially, starting with the later gestational ages (closer to the time of delivery) group first. Once the safety for this group is confirmed, groups of participants with earlier gestational ages will be enrolled.

Length of participation in this study will vary depending on gestational age at the time of enrollment, but each participant will have visits at study entry; Days 7, 14, and 28; 2 weeks after the last dose of the assigned gel; and once every 4 weeks until delivery. Participants who have used the gel within 24 hours of arriving at the hospital for delivery also will have a delivery visit. At most visits, participants will give a medical history; undergo blood and urine collection; and have a physical exam, including obstetric (OB) abdominal and pelvic exams. Participants also will report adverse events and complete an adherence assessment. If a participant has a delivery visit, blood will be collected from the umbilical cord and delivery and infant information will be collected. All participants will attend a follow-up study visit 30 days after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 45 years (inclusive) at screening, verified per site standard operating procedures (SOPs)
* At enrollment, singleton, viable pregnancy of gestational age within the limits for current group for enrollment
* Per participant report, sexually active, defined as having vaginal intercourse at least once in the 3 months prior to screening
* Able and willing to provide the following:

  * Written informed consent to be screened for and take part in the study
  * Adequate locator information, as defined in site SOPs
  * Adequate documentation of entry to antenatal care, as defined in site SOPs
  * Permission to contact and provision of adequate contact information for participant's antenatal care provider
  * Permission to obtain copies of antenatal care records More information on this criterion can be found in the protocol.
* HIV-uninfected based on testing performed by study staff at screening and enrollment (per algorithm in protocol)
* Per the clinical judgment of the Investigator of Record (IoR)/designee at enrollment, pelvic exam (including cervical exam) normal for estimated gestational age and parity
* Per the clinical judgment of the IoR/designee at enrollment, ultrasound results are complete, consistent with normal singleton intrauterine pregnancy, and provide an assessment of gestational age. More information on this criterion can be found in the protocol.
* Per participant mother report, willingness by the participant mother to receive information regarding and consider participation in MTN-016, a pregnancy registry study that collects additional information on pregnancy safety and the growth and development of babies up to 1 year of age
* At screening and enrollment, agrees not to participate in other research studies involving drugs, vaccines, medical devices, or vaginal products for the duration of study participation

Exclusion Criteria:

* Participant mother reported any of the following:

  * Prior exposure to gel or oral formulation of tenofovir (ever)
  * Known sensitivity to any component of the study products (ever)
  * Post-exposure prophylaxis (PEP) for HIV exposure within 6 months prior to enrollment
  * Participation in any research study involving drugs, medical devices, or vaginal products during the current pregnancy
  * Non-therapeutic injection drug use in the 12 months prior to screening
* By participant mother report, noted on antenatal record, or clinical evidence at the time of enrollment of any of the following in the current pregnancy:

  * Multiple gestation
  * Placenta previa
  * Cervical cerclage
  * Abnormal fetal anatomy (in the opinion of the IoR or designee)
  * Intrauterine growth restriction
  * Pre-existing or gestational diabetes
  * Hypertensive disorder of pregnancy
  * Treatment for preterm labor
* By participant mother report, or noted on review of medical record, any of the following in a previous pregnancy:

  * Intrauterine growth restriction
  * Gestational diabetes
  * Hypertensive disorder of pregnancy
  * Intrauterine fetal demise (estimated gestational age 20 weeks or greater)
  * Delivery prior to 37 0/7 weeks
* By participant mother report at screening or enrollment:

  * Intends to relocate away from the study site during the period of expected study visits
  * Plans to travel away from the study site during the expected study product dosing period, such that travel would preclude the completion of one or more scheduled study visits
  * Plans to deliver outside of a hospital. More information on this criterion can be found in the protocol.
* Currently breastfeeding
* As determined by the IoR/designee, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease, including active tuberculosis, or medication use that would make study participation unsafe. More information on this criterion can be found in the protocol.
* At enrollment, clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff). More information on this criterion can be found in the protocol.
* Has any of the following laboratory abnormalities during the screening period:

  * Hemoglobin value of Grade 3 or higher according to Division of AIDS (DAIDS) Toxicity Table
  * Platelet count less than 100,000 mm^3
  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 1.5 times the upper limit of normal
  * Serum creatinine greater than 1.0 mg/dL
  * Hepatitis B surface antigen (HBsAg) positivity
  * Urine dipstick positive for protein greater than or equal to 2
  * Urine dipstick positive for glucose greater than or equal to 2
  * Positive for malaria (at sites with capacity, where women are at risk and testing through antenatal care provider is not otherwise available)
  * More information on this criterion can be found in the protocol
* Grade 2 or higher Pap result (e.g., high-grade squamous intraepithelial lesion). More information on this criterion can be found in the protocol.
* Diagnosed with a sexually transmitted infection or reproductive tract infection requiring treatment, per current Centers for Disease Control and Prevention (CDC) or World Health Organization (WHO) guidelines, as applicable. More information on this criterion can be found in the protocol.
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Maternal outcomes: Grade 2 or higher adverse events (AEs) in select categories | Measured through participant's last study visit, which will occur 30 days after delivery
  Categories include: specific laboratory abnormalities, specific genital/pelvic signs/symptoms, and pregnancy complications
Neonatal outcomes (first 30 days of life): All serious adverse events (SAEs) | Measured through the 30 day follow-up visit

SECONDARY OUTCOMES:
Pharmacokinetics of tenofovir in mothers | Measured at Day 14 visit
  Blood samples will be collected pre- and post-tenfovoir dose to measure tenofovir levels and to estimate the maximum concentration (Cmax)
Self-reported product use captured through questionnaires | Measured through participant's last study visit, which will occur 30 days after delivery
Adherence to study gel as indicated by study drug levels in blood sample | Measured through participant's last study visit, which will occur 30 days after delivery
Adherence to study gel obtained by count of returned unused applicators | Measured through participant's last study visit, which will occur 30 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Beigi, MD, MSc, Study Chair — University of Pittsburgh; Bonus Makanani, MBBS, FCOG (SA), Study Chair — Kamuzu University of Health Sciences

REFERENCES:
- [Background] Abdool Karim Q, Abdool Karim SS, Frohlich JA, Grobler AC, Baxter C, Mansoor LE, Kharsany AB, Sibeko S, Mlisana KP, Omar Z, Gengiah TN, Maarschalk S, Arulappan N, Mlotshwa M, Morris L, Taylor D; CAPRISA 004 Trial Group. Effectiveness and safety of tenofovir gel, an antiretroviral microbicide, for the prevention of HIV infection in women. Science. 2010 Sep 3;329(5996):1168-74. doi: 10.1126/science.1193748. Epub 2010 Jul 19. PMID 20643915
- [Background] Nurutdinova D, Onen NF, Hayes E, Mondy K, Overton ET. Adverse effects of tenofovir use in HIV-infected pregnant women and their infants. Ann Pharmacother. 2008 Nov;42(11):1581-5. doi: 10.1345/aph.1L083. Epub 2008 Oct 28. PMID 18957630